Increasing Breast Cancer Screening in Chinese Immigrants PI: Dr. Lina Jandorf NCT05089292

Document Date: 2-24-2022


STUDY-20-01174 Form Version Date: January 15, 2022

#### **STUDY INFORMATION:**

Study Title: Increasing breast cancer screening in Chinese immigrants

Principal Investigator (Head Researcher): Lina Jandorf, MA

Physical Address: , New York, NY 10029

Mailing Address: One Gustave L. Levy Place Box 1077, NY, NY 10029

Phone: 212-659-5506

#### **SUMMARY OF THIS RESEARCH STUDY:**

In medicine, there are many unanswered questions. A research study is when scientists try to answer a question about something that we don't know enough about. Participation in a research study may or may not directly help you or others. Participation is entirely voluntary. It is completely up to you whether or not you take part. You can also change your mind at any time and it will not affect your ability to get medical care within the Mount Sinai Health System.

The purpose of this research study is to pilot test an education program with Chinese immigrant women to assess the feasibility and acceptability of an education program to improve mammogram screening utilization. The overall goal is to improve screening mammogram use in Chinese women in order to reduce disparities in cancer detection.

If you choose to participate, you will be asked to attend an education session on breast cancer screening and complete surveys on breast cancer screening history, knowledge, beliefs, and attitudes (as well as demographic data). There is no cost associated with your participation, and you will receive a \$30 gift card for your time and effort.

The main risks to you if you choose to participate are emotional discomfort associated with discussing breast cancer screening and breast cancer risk.

You may benefit from participating in this research by becoming more aware of the importance of screening mammograms for breast health.

If you are interested in learning more about this study, please continue to read below.

#### **PARTICIPATION IN THIS RESEARCH STUDY:**

This research study will be fully explained to you by a member of the study team. Feel free to ask all the questions you want before you make a decision about whether or not to participate. Any new information that develops during this research study that might make you change your mind about participating will be given to you promptly.

------FOR IRB USE ONLY-------



# 

STUDY-20-01174

Form Version Date: January 15, 2022

You may qualify to take part in this research study because you are: 1) 40 years of age or older, 2) female, 3) born in China, and 4) speak Cantonese, Mandarin, or English.

This research is being supported by a grant from the National Institutes of Health/National Institute on Minority Health and Health Disparities.

#### LENGTH OF TIME AND NUMBER OF PEOPLE EXPECTED TO PARTICIPATE:

Your participation in this research study is expected to last 60 minutes, including time for consenting and completing the surveys.

The number of people expected to take part in this research study is 72.

#### **DESCRIPTION OF WHAT'S INVOLVED:**

If you agree to participate in this research study, the following information describes what may be involved.

- Attend an education program on breast cancer risk and screening.
- Complete surveys asking you about your breast cancer screening history, knowledge, beliefs and attitudes. The survey will also ask you a few basic demographic questions (e.g., age, income, education level).
- This study will include one follow-up six months after attending the education program to assess breast cancer screening use.

The only research related ability that will need your involvement is completing the interviews. No invasive test (e.g., blood test, x-rays or other procedures) will be performed for the purposes of this research study. No drugs or device will be administered to you as part of this study.

# **USE OF YOUR DATA:**

The private information and/or data collected as part of this research will never be used or shared for future research, even if the identifiable information is removed.

#### YOUR RESPONSIBILITIES IF YOU TAKE PART IN THIS RESEARCH:

If you decide to take part in this research study, you will be responsible for the following things:

- Attending an education program
- Completing surveys

------FOR IRB USE ONLY------

ev 1.16.19

# 

STUDY-20-01174 Form Version Date: January 15, 2022

#### COSTS OR PAYMENTS THAT MAY RESULT FROM PARTICIPATION:

If you agree to take part in this research study, we will provide you with a \$30 gift card for your time and effort.

Tax law may require the Mount Sinai Finance Department to report the amount of payment you receive from Mount Sinai to the Internal Revenue Service (IRS) or other agencies, as applicable. Generally, this reporting would take place if you receive payments that equal \$600 or more from Mount Sinai in a calendar year. You would be responsible for the payment of any tax that may be due.

#### **POSSIBLE BENEFITS:**

It is important to know that you may not get any benefit from taking part in this research. Others may not benefit either. However, possible benefits may be learning more about breast density and its risks for breast cancer.

#### REASONABLY FORESEEABLE RISKS AND DISCOMFORTS:

- Psychological risks (for example, embarrassment, fear or stress). You might feel uncomfortable or distressed at answering some of the questions while completing the indepth telephone interviews.
- Risk of loss of private information; this risk always exists, but there are procedures in place to minimize the risk.
- You may have concerns about data security, privacy and confidentiality. Your name and other information that could directly identify you (such as address, date of birth) will be separated from study data and will never be placed into a scientific database.

### OTHER POSSIBLE OPTIONS TO CONSIDER:

You may decide not to take part in this research study without any penalty. The choice is totally up to you.

#### IN CASE OF INJURY DURING THIS RESEARCH STUDY:

If you believe that you have suffered an injury related to this research as a participant in this study, you should contact the Principal Investigator.

#### **ENDING PARTICIPATION IN THE RESEARCH STUDY:**

You may stop taking part in this research study at any time without any penalty. This will not affect your ability to receive medical care at any of the Mount Sinai Health System hospitals or to receive any benefits to which you are otherwise entitled.

-----FOR IRB USE ONLY------

ev 1.16.19

# 

#### STUDY-20-01174

Form Version Date: January 15, 2022

If you decide to stop being in the research study, please contact the Principal Investigator or the research staff.

If you decide you don't want your data to be used for research anymore, you can contact the researcher and ask to have your data removed. Data that have already been used will not be affected by your decision. Any data that are still linked to your identity by a code the researcher has will be withdrawn.

<u>Withdrawal without your consent</u>: The study doctor, the sponsor or the institution may stop your involvement in this research study at any time without your consent. This may be because the research study is being stopped, the instructions of the study team have not been followed, the investigator believes it is in your best interest, or for any other reason. If data has been stored as part of the research study, they too can be destroyed without your consent.

#### **CONTACT INFORMATION:**

If you have any questions, concerns, or complaints at any time about this research, or you think the research has harmed you, please contact the office of the research team and/or the Principal Investigator, Lina Jandorf at phone number: 212-659-5506.

This research has been reviewed and approved by an Institutional Review Board. You may reach a representative of the Program for Protection of Human Subjects at the Icahn School of Medicine at Mount Sinai at telephone number (212) 824-8200 during standard work hours for any of the reasons listed below. This office will direct your call to the right person within the Mount Sinai Health System:

- Your questions, concerns, or complaints are not being answered by the research team.
- You cannot reach the research team.
- You are not comfortable talking to the research team.
- You have questions about your rights as a research subject.
- You want to get information or provide input about this research.

# **DISCLOSURE OF FINANCIAL INTERESTS:**

Sometimes, physicians/researchers receive payments for consulting or similar work performed for industry. Effective September 2014 Mount Sinai reviews only payments to an individual totaling more than \$5,000 a year per entity when determining potential conflicts of interest. If you have questions regarding industry relationships, we encourage you to talk your physician/researcher or visit our website at http://icahn.mssm.edu/ where Mount Sinai publicly discloses the industry relationships of our faculty.

#### **MAINTAINING CONFIDENTIALITY - HIPAA AUTHORIZATION:**

As you take part in this research project, it will be necessary for the research team and others to use and share some of your private protected health information. Consistent with the federal Health

ev 1.16.19

-----FOR IRB USE ONLY------

# THE MOUNT SINAI HEALTH SYSTEM CONSENT FORM TO VOLUNTEER IN A RESEARCH STUDY AND AUTHORIZATION FOR USE AND DISCLOSURE OF MEDICAL INFORMATION

**Icahn School of Medicine at Mount Sinai** 

# 

#### STUDY-20-01174

Form Version Date: January 15, 2022

Insurance Portability and Accountability Act (HIPAA), we are asking your permission to receive, use and share that information.

What protected health information is collected and used in this study, and might also be shared with others?

As part of this research project, the research team at the hospital(s) involved in the research will collect your name, address, telephone, or email.

During the study the researchers will gather information by:

- completing the in-depth interview explained in the description section of this consent

## Why is your protected health information being used?

Your personal contact information is important to be able to contact you during the study. Your health information and the results of any tests and procedures being collected as part of this research study will be used for the purpose of this study as explained earlier in this consent form. The results of this study could be published or presented at scientific meetings, lectures, or other events, but would not include any information that would let others know who you are, unless you give separate permission to do so.

The research team and other authorized members of The Mount Sinai Health System ("Mount Sinai") workforce may use and share your information to ensure that the research meets legal, institutional or accreditation requirements. For example, the School's Program for the Protection of Human Subjects is responsible for overseeing research on human subjects, and may need to see your information. If you receive any payments for taking part in this study, the Mount Sinai Finance Department may need your name, address, social security number, payment amount, and related information for tax reporting purposes. If the research team uncovers abuse, neglect, or reportable diseases, this information may be disclosed to appropriate authorities.

#### Who, outside Mount Sinai, might receive your protected health information?

As part of the study, the Principal Investigator, study team and others in the Mount Sinai workforce may disclose your protected health information, including the results of the research study and procedures, to the following people or organizations: (It is possible that there may be changes to the list during this research study; you may request an up-to-date list at any time by contacting the Principal Investigator.)

- The United States Department of Health and Human Services and the Office of Human Research Protection.

In all disclosures outside of Mount Sinai, you will not be identified by name, address, telephone number, or any other direct personal identifier unless disclosure of the direct identifier is required by law. Some records and information disclosed may be identified with a unique code number. The Principal Investigator will ensure that the key to the code will be kept in a locked file, or will be securely stored electronically. The code will not be used to link the information back to you without your permission, unless the law requires it, or rarely if the Institutional Review Board allows it after determining that there would be minimal risk to your privacy. It is possible that a sponsor or their representatives, a data

------FOR IRB USE ONLY-------ev 1.16.19



# THE MOUNT SINAI HEALTH SYSTEM CONSENT FORM TO VOLUNTEER IN A RESEARCH STUDY AND AUTHORIZATION FOR USE AND DISCLOSURE OF MEDICAL INFORMATION

**Icahn School of Medicine at Mount Sinai** 

# 

Form Version Date: January 15, 2022

#### STUDY-20-01174

coordinating office, a contract research organization, may come to inspect your records. Even if those records are identifiable when inspected, the information leaving the institution will be stripped of direct identifiers. Additionally, when applicable, the monitors, auditors, the IRB, the Office of Human Subjects Protection (OHRP) of the Department of Health and Human Services as well as the Food and Drug Administration (FDA) will be granted direct access to your medical records for verification of the research procedures and data. OHRP and FDA are authorized to remove information with identifiers if necessary to complete their task. By signing this document you are authorizing this access. We may publish the results of this research. However, we will keep your name and other identifying information confidential.

For how long will Mount Sinai be able to use or disclose your protected health information? Your authorization for use of your protected health information for this specific study does not expire.

### Will you be able to access your records?

During your participation in this study, you will have access to your medical record and any study information that is part of that record. The investigator is not required to release to you research information that is not part of your medical record.

# Do you need to give us permission to obtain, use or share your health information?

NO! If you decide not to let us obtain, use or share your health information you should not sign this form, and you will not be allowed to volunteer in the research study. If you do not sign, it will not affect your treatment, payment or enrollment in any health plans or affect your eligibility for benefits.

# Can you change your mind?

You may withdraw your permission for the use and disclosure of any of your protected information for research, but you must do so in writing to the Principal Investigator at the address on the first page. Even if you withdraw your permission, the Principal Investigator for the research study may still use your protected information that was already collected if that information is necessary to complete the study. Your health information may still be used or shared after you withdraw your authorization if you should have an adverse event (a bad effect) from being in the study. If you withdraw your permission to use your protected health information for research that means you will also be withdrawn from the research study, but standard medical care and any other benefits to which you are entitled will not be affected. You can also tell us you want to withdraw from the research study at any time without canceling the Authorization to use your data.

It is important for you to understand that once information is disclosed to others outside Mount Sinai, the information may be re-disclosed and will no longer be covered by the federal privacy protection regulations. However, even if your information will no longer be protected by federal regulations, where possible, Mount Sinai has entered into agreements with those who will receive your information to continue to protect your confidentiality.

If as part of this research project your medical records are being reviewed, or a medical history is being taken, it is possible that HIV-related information may be revealed to the researchers. If that is the case,



-----FOR IRB USE ONLY------

# 

STUDY-20-01174

Form Version Date: January 15, 2022

the following information concerns you. If this research does not involve any review of medical records or questions about your medical history or conditions, then the following section may be ignored.

# **Notice Concerning HIV-Related Information**

If you are authorizing the release of HIV-related information, you should be aware that the recipient(s) is (are) prohibited from re-disclosing any HIV-related information without your authorization unless permitted to do so under federal or state law. You also have a right to request a list of people who may receive or use your HIV-related information without authorization. If you experience discrimination because of the release or disclosure of HIV-related information, you may contact the New York State Division of Human Rights at (888) 392-3644 or the New York City Commission on Human Rights at (212) 306-5070. These agencies are responsible for protecting your rights.

------FOR IRB USE ONLY------



# 

STUDY-20-01174 Form Version Date: January 15, 2022

| | n information. A signed and dated copy | research and to the use and will be given to you. |
|---|---|---|
| Signature of subject | Printed Name of Subject | Date |
| PERSON EXPLAINING STUDY A | AND OBTAINING CONSENT: | |
| Signature of consent delegate | Printed Name of consent delegate | Date |
| | observe the consent process, it should<br>te, visually impaired, or this documer | |
| | hat the information in the consent doc<br>ned to, and apparently understood by, | |
| information was accurately explai | | |
| information was accurately explai was freely given by the subject. | ned to, and apparently understood by, | the subject, and that consent |
| information was accurately explai was freely given by the subject. | ned to, and apparently understood by, | the subject, and that consent |